CLINICAL TRIAL: NCT01067053
Title: A Non Randomized Phase II Trial to Assess Efficacy and Safety of Bevacizumab, Capecitabine and Oxaliplatin as First Line Treatment for Elderly Patients With Metastatic Colorectal Adenocarcinoma, Suitable for Polychemotherapy Treatment
Brief Title: Efficacy/Safety Study of Bevacizumab,Capecitabine,Oxaliplatin to Metastatic Colorectal Adenocarcinoma Elderly Patients.
Acronym: BECOX
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Grupo Espanol Multidisciplinario del Cancer Digestivo (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEMCAD-0901
Record Dates: First submitted 2010-01-21; First posted 2010-02-11 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2014-01

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Bevacizumab; Capecitabine; Oxaliplatin; Metastatic colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab; Capecitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- bevacizumab, capecitabine, oxaliplatin (Experimental): 6 cycles (3 weeks each one) of:
  * bevacizumab: 7,5 mg/kg (iv), 1st day of each cycle.
  * capecitabine: 1000 mg/m2 bid, oral. Days: 1-14 every three weeks.
  * oxaliplatin: 130/mg/m2(iv),1st day of each cycle.
  After the first 6 cycles of treatment, continuing only with bevacizumab and capecitabine
  Interventions: Drug: bevacizumab, capecitabine, oxaliplatin

INTERVENTIONS:
Drug: bevacizumab, capecitabine, oxaliplatin — 6 cycles (3 weeks each one) of:
  * bevacizumab: 7,5 mg/kg (iv), 1st day of each cycle.
  * capecitabine: 1000 mg/m2 bid, oral. Days: 1-14 every three weeks.
  * oxaliplatin: 130/mg/m2(iv),1st day of each cycle.
  After the first 6 cycles of treatment, continuing only with bevacizumab and capecitabine
  Other Names: bevacizumab (Avastin®); capecitabine (Xeloda®); oxaliplatin

SUMMARY:
The purpose of this study is to determine whether bevacizumab, capecitabine and oxaliplatin are an effective and safe first line of treatment for elderly patients with metastatic colorectal adenocarcinoma.

DETAILED DESCRIPTION:
The efficacy will be determined by objective response rate following RECIST criteria.

In several clinical trials with Bevacizumab, there has been demonstrated that elderly patients benefits as well as the younger of a combination therapy with chemotherapy plus Bevacizumab, but these results have come from subgroup analyses of trials not specifically design to test the effect of these combinations on the elderly. This clinical trial is specific only for elderly patients and we expect to confirm the benefits demonstrated in other clinical trials where the elderly patients were a number reduced.

This clinical trial includes 3 substudies:

- Assessment of tumor response of CRC liver metastases to treatment with Avastin in combination with Capecitabine and Oxaliplatin as first line treatment by dynamic ultrasound contrast.

Main objective: Assess the performance of dynamic contrast ultrasonography (CEUS, Contrast Enhanced UltraSound) with quantification of tumor perfusion in the evaluation of tumor response of liver metastases of colorectal carcinoma to treatment with Avastin in combination with Capecitabine and Oxaliplatin.

-Evaluation of the antiangiogenic activity of bevacizumab combined with oxaliplatin and capecitabine in first line treatment using MDCT perfusion studies in liver metastases of colorectal cancer in patients over 70 years.

Main objective:Determine whether the observed changes in perfusion CT studies performed at 2 weeks of starting treatment compared to baseline are significant predictors of free time to disease progression in patients in the trial and defined as the time since the start of treatment until objective progressive disease by RECIST criteria.

-Characterization of resistance to bevacizumab in colon cancer in elderly patients.

Main objective: To evaluate the involvement of serum markers and markers in the primary tumor in the resistance to bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* ECOG 0-1.
* Age ≥ 70 years.
* Histologically confirmed carcinoma of the colon and/or rectum.
* Metastatic disease non suitable for radical surgery.
* At least one measurable metastatic lesion (as per RECIST criteria). The index lesion must not be in a previously irradiated area.
* Non prior chemotherapy for metastatic disease. Adjuvant (or neo-adjuvant for rectal cancer patients) chemotherapy allowed if completed ≥ 12 months before inclusion.
* Life expectancy more than 3 months.
* Adequate renal function: creatinine ≤ 1.5 x UL and calculated creatinine clearance ≥ 30 mL/min.
* Adequate level function: AST and ALT ≤ 2.5 x UL (≤ 5 x UL if liver metastases), bilirubin ≤ 1.5 x UL.
* Adequate haematological function: Hb ≥ 9 gr/dl, neutrophils ≥ 1,5 x 109 /l and platelets ≥ 100000 x 109/l.
* Urine dipstick for proteinuria < 2+. If urine dipstick is ≥ 2+, 24 hour urine must demonstrate ≤ 1 g of protein in 24 hours.
* No clinical evidence or history of metastatic CNS disease.
* No prior Bevacizumab treatment.

Exclusion Criteria:

* Patients who previously received bevacizumab.
* Prior chemotherapeutic treatment for metastatic CRC.
* Prior treatment with monoclonal antibodies.
* Clinical evidence of brain metastases or history or evidence upon physical examination of CNS disease unless adequately treated.
* Past or current history (within the last 5 years prior to treatment start) of other malignancies except metastatic colorectal cancer (Patients with curatively treated basal and squamous cell carcinoma of the skin or in situ carcinoma of the cervix are eligible).
* Clinically significant cardiovascular disease, for example CVA (≤ 6 months before treatment start), myocardial infarction (≤ 6 months before treatment start), unstable angina, NYHA ≥ grade 2, CHF, arrhythmia requiring medication, or uncontrolled hypertension.
* Intestinal occlusion/subocclusion.
* Chronic diarrhea.
* Treatment with any other investigational agent, or participation in another clinical trial within 30 days prior to entering this study.
* Known hypersensitivity to any of the study drugs.
* Current or recent (within 10 days of first dose of study treatment) daily use of aspirin (> 325 mg/day) or other NSAID.
* Current or recent (within 10 days prior to study treatment start) use of full-dose oral or parenteral anticoagulants or thrombolytic agent for therapeutic (as opposed to prophylactic) purposes. Patients receiving (or considered candidate to receive) anticoagulants agents as prophylaxis of cardiovascular risk, should continue (or start) the appropriate treatment at study entry.
* History of venous thromboembolic or haemorrhagic events within 6 months prior to treatment.
* Patients with previous of arterial thromboembolic event.
* Evidence of bleeding diathesis or coagulopathy.
* Serious, non healing wound, ulcer, or bone fracture.
* Major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to treatment, or anticipation of the need for major surgery during the course of the study.
* Evidence of any other disease, metabolic dysfunction, physical examination finding or laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or puts the patient at high risk for treatment-related complications.
* Patients of childbearing potential not willing to use effective means of contraception.
* Positive HIV serology.
* Known addiction to alcohol or other drugs.
* Patients included in other clinical trial

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-11 (Actual); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Time to progression | 3 years

SECONDARY OUTCOMES:
Overall survival | 3 years
Objective response rate following Response Evaluation Criteria In Solid Tumors (RECIST) criteria | 3 years
Overall response rate | 3 years
Number of treatment cycles administered | 3 years
Number of patients who have required dose reductions of either drug | 3 years
Safety of treatment according to the number of adverse events reported | 3 yeras

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Feliu Batlle, MD, Study Chair — Grupo Español Multidisciplinario de Cáncer Digestivo
Locations (15):
- Spain (15):
  - Hospital Clinic i Provincial, Barcelona, Barcelona
  - Hospital de L´Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Hospital General Yagüe, Burgos, Burgos
  - Hospital de Gran Canaria Doctor Negrin, Las Palmas de Gran Canaria, Las Palmas
  - Hospital Arnau de Vilanova, Lleida, Lérida
  - Hospital Universitario la Paz, Madrid, Madrid
  - Hospital Quirón de Madrid, Madrid, Madrid
  - Hospital Infanta Sofía, San Sebastián de los Reyes, Madrid
  - Hospital Morales Meseguer, Murcia, Murcia
  - Hospital de Navarra, Pamplona, Navarre
  - Hospital La Fe de Valencia, Valencia, Valencia
  - Hospital General de Valencia, Valencia, Valencia
  - Hospital Doctor Peset, Valencia, Valencia
  - Hospital Lluis Alcanyis, Xàtiva, Valencia
  - Hospital Xeral Cies de Vigo, Vigo, Vigo